CLINICAL TRIAL: NCT06645262
Title: First-degree Ankle Sprains
Status: Recruiting | Type: Observational
Sponsor: Rehabilitation Centre Zivot (Other)
Responsible Party: Principal Investigator, Darko Bilic, Director, Rehabilitation Centre Zivot
Other Study IDs: A2024
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Ankle Sprain 1St Degree
Keywords: ankle sprain; Bowen technique
MeSH Terms: conditions — Ankle Injuries | interventions — Cryotherapy; Braces

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: In this group, the intervention will consist of cryotherapy, therapeutic exercises, the use of braces, and the Bowen technique.
  Interventions: Other: Cryotherapy
- Control Group: In this group, the intervention will consist of cryotherapy, therapeutic exercises, the use of braces, and manual massage.
  Interventions: Other: Cryotherapy

INTERVENTIONS:
Other: Cryotherapy — cryotherapy, therapeutic exercises, the use of braces, and the Bowen technique.
  Other Names: cryotheraphy; braces; Bowen technique

SUMMARY:
Grade I ankle sprains are common, especially among athletes, women, teenagers, and physically active individuals. While over a million cases are reported annually, this represents only half of the total occurrences. These injuries can lead to complications like chronic ankle instability or osteoarthritis. Treatment often involves conservative methods, including the PRICEMMS protocol (protection, rest, ice, compression, elevation, modalities, medication, and support), while surgery is reserved for severe cases. Therapeutic exercises and rehabilitation play a key role in recovery. The Bowen technique, effective for other musculoskeletal issues, has not yet been extensively studied for Grade I ankle sprains.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with Grade I acute ankle sprain confirmed by a specialist physician in radiology,
* Age of participants ≥ 18 years,
* Individuals of both sexes

Exclusion Criteria:

* Recurrent ankle injury,
* Acute ankle sprains of Grade II and III,
* Presence of other physical and/or mental health issues.

Min Age: 18 Weeks | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The sample is a convenience sample and will include individuals diagnosed with Grade I acute ankle sprain who present for examination at the specified institutions. After a proper diagnosis, confirmation of inclusion in the study, and signed ethical consent for participation in the research, randomization of participants will be conducted using an electronic number generator on the website www.randomizer.org/form:htm.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Subjective assessment of pain intensity | 3 weeks
  Measured on a numerical scale ranging from 0 to 10

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation Centre Život, Mostar, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Undecided